CLINICAL TRIAL: NCT03132896
Title: Re-Evaluation of Systemic Early Neuromuscular Blockade and Transthoracic Ultrasound Assessment of the Diaphragm
Acronym: ROSETTA
Status: Withdrawn | Type: Observational
Why Stopped: Investigational device no longer has Health Canada approval.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 16-6360
Record Dates: First submitted 2017-04-19; First posted 2017-04-28 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2018-07

CONDITIONS: Acute Respiratory Distress Syndrome; Diaphragm Injury; Neuromuscular Blockade
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with moderate or severe ARDS

SUMMARY:
ROSETTA is a multi-centre study evaluating the time course of diaphragm thickness and function following exposure to neuromuscular blockade or control in patients with acute respiratory distress. ROSETTA is an ancillary study to the Re-evaluation of Systemic Early Neuromuscular Blockade (ROSE) trial (NCT02509078). It is designed to (1) test the feasibility of a multi-center evaluation of the diaphragm structure and function by ultrasound during mechanical ventilation and (2) determine whether neuromuscular blockade accelerates atrophy and dysfunction of the diaphragm in patients with acute respiratory distress syndrome (ARDS).

DETAILED DESCRIPTION:
A growing body of evidence strongly suggests that mechanical ventilation injures the respiratory muscles, particularly the diaphragm. Due to the deleterious effects of diaphragm inactivity on diaphragm function, there are important concerns about the risk of diaphragm weakness and difficult liberation from mechanical ventilation following neuromuscular blockade. Sonographic measurements of diaphragm thickness provide a potentially useful window for studying diaphragm injury and function during mechanical ventilation.

Patients enrolled in the ROSE trial (randomizing patients with moderate-severe acute respiratory distress syndrome to receive neuromuscular blockade or control for 2 days) will be eligible for participation in this study. Study patients will undergo regular diaphragm ultrasound to assess diaphragm thickness and activity during the first week of the study. Diaphragm function will be assessed by ultrasound on study days 7, 14, 21, and 28.

ROSETTA is designed to:

1. Test the feasibility of a multi-center evaluation of the diaphragm structure and function by ultrasound during mechanical ventilation;
2. Determine whether neuromuscular blockade accelerates atrophy and dysfunction of the diaphragm in patients with acute respiratory distress syndrome; and
3. Evaluate whether patients with greater diaphragm dysfunction exhibit worse functional outcomes compared to patients without diaphragm dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Patients enrolled in the ROSE PETAL trial (adult patients with moderate-severe acute respiratory distress syndrome who have received invasive mechanical ventilation for less than 5 days)

Exclusion Criteria:

1. Patients expected to be extubated within 24 hours of screening for eligibility
2. Patients with a contraindication to chest ultrasonography (chest tubes inserted over right lower chest wall; chest wall trauma)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe acute respiratory distress syndrome (ARDS) who consent to the ROSE trial will be invited to participate in the ROSETTA study.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Study feasibility - number of participating centers | Through study completion, an average of 18 months
  The number of centers that participate in the study
Study feasibility - number of trained sonographers in study | Through study completion, an average of 18 months
  The number of trained sonographers who collect measurements with ultrasound in the study
Study feasibility - enrolment rate | Through study completion, an average of 18 months
  Percentage of potentially eligible patients in ROSE trial who are enrolled in ROSETTA
Study feasibility - measurement acquisition rate | Through study completion, an average of 18 months
  Percentage of scheduled study measurements that are actually collected

SECONDARY OUTCOMES:
Diaphragm function | Study day 7
  Maximal diaphragm thickening fraction
Changes in diaphragm thickness over time with or without neuromuscular blockade | First week of study

CONTACTS AND LOCATIONS:
Overall Officials: Ewan C Goligher, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (6):
- United States (6):
  - Brigham and Women's Health, Boston, Massachusetts
  - Baystate Health, Springfield, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes